CLINICAL TRIAL: NCT05780372
Title: Reduced Volume of Neck Prophylactic Irradiation in Nasopharyngeal Carcinoma: a Multi-center, Non-inferiority, Open-label, Randomized Controlled Phase III Clinical Trial
Brief Title: Reduced Volume of Neck Prophylactic Irradiation in Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangxi Provincial Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Chongqing University Cancer Hospital (Other); Dongguan People's Hospital (Other Government); LiuZhou People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Chong, Doctor, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reduced CTV in NPC
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma; Radiotherapy; Complications
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced CTVn2 (Experimental): Patients will receive the reduced neck prophylactic irradiation, only the level of positive lymph nodes and its next level.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Chemotherapy
- Conventional CTVn2 (Active Comparator): Patients will receive the conventional neck prophylactic irradiation, as suggested by the international guideline.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — All target volumes will be outlined slice by slice on the axial contrast-enhanced CT with MR fusion images in the treatment planning system. The target volumes are defined in accordance with the International Commission on Radiation Units and Measurements Reports 83. The prescribed dose is 70-72 Gy to PTVp (Planning target volume of the primary tumor), 64-70 Gy to PTVn (Planning target volume of the lymph node),60- 64Gy to PTV1 (High-risk planning target volume), and 54-58 Gy to PTV2 (Low-risk planning target volume) in 30-32 fractions. The details of dose limits for organs at risk are based on the study 0225 from The Radiation Therapy Oncology Group (RTOG 0225).
  Other Names: IMRT
Drug: Chemotherapy — Chemotherapy will be arranged by the physician-in-charge according to the NCCN guideline, patient's stage and physical condition.

SUMMARY:
This is a multi-center, non-inferiority, open-label, randomized controlled phase III clinical trial in primary diagnosed nasopharyngeal carcinoma (NPC) patients without distant metastasis. The purpose of this study is to evaluate the efficacy of reduced neck prophylactic radiotherapy versus conventional neck prophylactic radiotherapy, and compare the radiotherapy-related adverse events and quality of life in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal non-keratinizing carcinoma (WHO II/III);
* All genders, range from 18-70 years old;
* ECOG score 0-1;
* Clinical stage I-IVa (AJCC/UICC 8th);
* Not received radiotherapy, chemotherapy and other anti-tumor treatment (including immunotherapy);
* No contraindications to chemotherapy or radiotherapy;
* Adequate organ function: white blood cell count ≥ 4×109/L, neutrophile granulocyte count ≥ 1.5×109/L, hemoglobin ≥ 9g/L, platelet count ≥ 100×109/L; alanine aminotransferase or aspartate aminotransferase < 2.5×upper limit of normal; blood urea nitrogen or creatinine ≤ 1.5×upper limit of normal or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* Sign the consent form.

Exclusion Criteria:

* Neck lymph nodes exist skipping metastasis;
* Distant metastases;
* Keratinized squamous cell carcinoma or basal cell like squamous cell carcinoma;
* Have or are suffering from other malignant tumors;
* Participating in other clinical trials;
* Pregnancy or lactation;
* Have uncontrolled cardiovascular disease;
* Severe complication, eg, uncontrolled hypertension;
* Mental disorder;
* Drug or alcohol addition;
* Do not have full capacity for civil acts.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Regional recurrence-free survival | 3 years
  From the date of randomization to regional recurrence or any death

SECONDARY OUTCOMES:
Overall survival | 3 years
  From the date of randomization to any death, with patients unavailable for follow-up censored at the date of last follow-up
Local recurrence-free survival | 3 years
  From the date of randomization to local recurrence or any death
Distant metastasis-free survival | 3 years
  From the date of randomization to distant metastasis or any death
Progression free survival | 3 years
  From the date of randomization to local or regional recurrence, distant metastasis or any death
Acute toxicities | From the start of treatment until 3 months post treatment
  Assessed with CTCAE v5.0
Late toxicities | 3 years post treatment
  Assessed with RTOG/EORTC
Quality of life score | During treatment and 3 years post treatment
  Assessed with EORTC-Quality of life questionnaire-C30 version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, MD PhD, Principal Investigator — Sun Yat-sen University
Locations (7):
- China (7):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Dongguan People Hospital, Dongguan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Jiangxi Cancer Hospital of Nanchang University, Nanchang, Jiangxi
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn